CLINICAL TRIAL: NCT01892111
Title: Structured Exerise Training in Infertile Obese Patients Treated With Assisted Reproductive Techniques: a Randomized Controlled Trial
Brief Title: Physical Activity and ARTs
Acronym: SETART
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2013
Record Dates: First submitted 2013-06-28; First posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-06

CONDITIONS: Infertility; Obesity; Stable BMI
Keywords: SET; infertility; IVF/ICSI; pregnancy
MeSH Terms: conditions — Infertility; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- structured exercise program (SET) (Experimental): SET one month before and during ARTs. IVF/ICSI procedure.
  Interventions: Other: Structured exercise program.
- no intervention (No Intervention): IVF/ICSI procedure.

INTERVENTIONS:
Other: Structured exercise program.
  Arms: structured exercise program (SET)

SUMMARY:
Obese women experience increased infertility rate and longer time to conception showing lower pregnancy and live-birth rates both in natural and assisted conceptions. Body weight loss improves not only spontaneous pregnancy rates but also those of assisted reproductive techniques (ARTs). Almost all studies refer to body weight loss due to lifestyle intervention programs consisting in hypocaloric diet and increased physical activity, whereas very little is known about the specific effects of physical activity alone on human reproduction.

In a previous retrospective study, we demonstrated that physical activity enhances the reproductive performance of obese infertile patients who receive in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI) cycles, regardless of body weight loss.

The aim of this randomized controlled trial (RCT) will be to evaluate if a structured exercise program improve the effectiveness of ARTs.

DETAILED DESCRIPTION:
Women with primary infertility scheduled to an IVF/ICSI procedure, obese and with a stable BMI will be randomized to receive a structured exercise program or nothing.

Patients will undergo a gonadotropin ovarian hyperstimulation for standard IVF/ICSI procedure.

clinical and biological data will be evaluated in each subject.

ELIGIBILITY:
Inclusion Criteria:

* infertility
* obesity
* stable BMI
* schedule for ARTs

Exclusion Criteria:

* use of cryopreserved embryos
* any changes in diet and physical activity
* tobacco smoking
* drug use
* alcohol abuse
* uterine diseases
* previous pelvic surgery
* major medical diseases
* clinical history of (or suspicion of) endometriosis, antiphospholipid antibody syndrome, recurrent miscarriage
* obese partner
* severe sperm pathology

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate. | 4 months

SECONDARY OUTCOMES:
stimulation lenght and dose | 1 month
cancellation rate | 1 months
implantation rate | 1 month
OHSS rate | 1 month
embryo transferred | 1 month
miscarriage rate | 4 months
multiple pregnancy rate | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Gynecology & Obstetrics - Arcispedale S. Maria Nuova of Reggio Emilia, IRCCS, University of Modena and Reggio Emilia, Reggio Emilia, Italy

REFERENCES:
- [Background] Palomba S, Falbo A, Giallauria F, Russo T, Rocca M, Tolino A, Zullo F, Orio F. Six weeks of structured exercise training and hypocaloric diet increases the probability of ovulation after clomiphene citrate in overweight and obese patients with polycystic ovary syndrome: a randomized controlled trial. Hum Reprod. 2010 Nov;25(11):2783-91. doi: 10.1093/humrep/deq254. Epub 2010 Sep 21. PMID 20858697
- [Background] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291